CLINICAL TRIAL: NCT02407977
Title: Real Time In-Vivo Body Surface Dosimetry for External Beam Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00061601
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cancer of the Gastrointestinal, Genitourinary or Gynecologic Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Novel nano-scintillatorfiber-optic dosimeter ( nanoFOD) — This is an observational study whose purpose is to determine the feasibility of using a novel nano-scintillator fiber-optic dosimeter ( nanoFOD) for real time dosimetric monitoring of external beam radiotherapy.
  Other Names: nanoFOD

SUMMARY:
This is an observational study. This protocol will determine the feasibility of using a novel nano-material based fiber-optic dosimeter (nanoFOD) device, with dimensions less than 1 mm wide, to measure real-time, pin-point, in-vivo radiation dose given during external beam delivery of radiation therapy treatments.This new protocol is similiar in design to Pro00050297 with the significant difference being the monitoring will be performed during external baem radiotherapy.

DETAILED DESCRIPTION:
The device is currently in use in an ongoing IRB approved protocol Pro00050297 "Real Time In-Vivo Dosimetry For Gynecologic Brachytherapy". Brachytherapy is an integral part of the management of many gynecological cancers, which uses radioactive isotopes to deliver radiation treatment in close proximity to the target. The protocol uses the device in the setting of gynecologic brachytherapy to monitor real time doses, with a primary endpoint of feasibility and accuracy. Accrual is ongoing, however, the device has initially given consistent results, within 3% of the expected values. This initial experience is intentionally designed with the simplest geometry and positioning. This protocol has a similar design to the initial brachytherapy trial, but with the significant difference that the monitoring will be performed during external beam radiotherapy. Calibration procedures are different in this scenario, and the considerations of when and where dose monitoring will be useful are distinct from these considerations in brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented neoplasm of the pelvis (including gynecologic, gastrointestinal, and genitourinary origin).
* Planned external beam radiotherapy as part of standard of care treatment
* The radiotherapy plan involves the body surface
* Age > 18 years
* Able to provide and execute informed consent

Exclusion Criteria:

* Allergy or previous intolerance of skin adhesives
* Any clinical scenario in which the nanoFOD placement or reading would compromise the treatment efficacy, or endanger the patient in any way.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with histologically documented neoplasm of the pelvis (including gynecologic, gastrointestinal, and genitourinary origin).
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Dosimetric accuracy of the device with reference to a commercially available dosimeter | 24 months

SECONDARY OUTCOMES:
Feasibility of clinical application of the nanaoFOD for dosimetric monitoring of external beam radiotherapy. | 24 months
  Feasibility in this context will mean ease of clinical use (subjective) and lack of device failures.

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Chino, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medica Center, Durham, North Carolina, United States